CLINICAL TRIAL: NCT04942938
Title: A Pilot Study of Neubie, a Direct Current Electrical Stimulation Device, to Inhibit Lower Extremity Spasticity Levels and Normalize Muscle Functional Use During Transfers and Ambulation in Individuals With Multiple Sclerosis
Brief Title: Impact of Direct Current Electrical Stimulation on Spasticity Levels and Functional Muscle Use in MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CommonSpirit Health (Other)
Collaborators: NeuFit - Neurological Fitness and Education (Industry)
Responsible Party: Principal Investigator, Courtney Ellerbusch, Physical Therapist, CommonSpirit Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1643900-2
Record Dates: First submitted 2021-06-01; First posted 2021-06-29 (Actual); Results first posted 2025-04-18 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: This will be a pilot study using a series of 4-6 case studies for 4-6 participants. All studies will be completed entirely from the subject's home with CSHRI IRB oversight.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Neubie Treatment (Experimental): Participants in this study will participate in intervention treatment with the Neubie for 6 weeks. Outcome measures objective and subjective will be collected at the beginning and end of the study. The treatments will include:
  1. Manual activations to underactive, spastic or limited in sensory muscles/regions
  2. Neubie Mapping mode scanning process to scan for 1) spots that stimulate movement they couldn't do before per initial assessment, 2) spots that allow movement which is a greater range than available before per initial assessment, 3) spots that lead to decreased spasticity, and 4) diminished sensation areas - drive signal to increase sensory nerves and become metabolically active.
  3. Train using physical therapy exercises with Neubie in training mode and Hz current adjusted for tolerance (perceived 7/10) and ability to work through or decrease spasticity in (500 Hz) in the areas which show spasticity, contraction, are dead/diminished sensation, and hot spots.
  Interventions: Device: Neubie

INTERVENTIONS:
Device: Neubie — The Neubie is a direct current neuromuscular electrical stimulation device. This system uses an exponential wave pattern to mimic the natural pattern neurologically to lengthen fibers of the sarcomere and engage force velocity of muscle with minimized protective co-contraction of nearby muscle groups. The golgi tendon and muscle spindles code for joint position and muscle/tendon stretch with 66% of fibers being intrafusal. Impacting these structures has direct impact on reticulospinal tract fibers and proprioceptive central fibers modulation of levels of spasticity. The Neubie direct current is designed to improve positioning of these stretch receptors.

SUMMARY:
In an individual with MS the central nervous system (CNS) is over-protective and causes the threshold for stretch reflex and muscle tightness to be set lower than normal. This inhibits normal movement and causes abnormalities in posture, stiffness and at times joint contractures. In this pilot study we hope to assess the ability for the direct current of Neubie, which creates mechanoreceptor inputs and lengthening at the sarcomere level of muscle and joints in the spine and lower extremity, to alter the proprioceptive peripheral nervous system (PNS) at muscle spindle and GTO level with a change in CNS over-guarding during the treatment and after the treatment. If the investigators are able to create normalized stretch and muscle tension at the PNS level, it may be possible to create temporary or sustained CNS level changes. This would allow the amount of stretch and tension at the PNS level to be normalized and possibly reduce spasticity. If this theory is accurate, the investigators may be able to increase access to normalized movement, strength and functional ability in individuals with neuro-compromise.

DETAILED DESCRIPTION:
Approximately 66%6 to 84% of individuals with multiple sclerosis experience various levels of debilitating spasticity limiting freedom of movement at ankles, knees and hips causing deficits in ambulation, weakness from disuse of muscles not accessible due to spasticity. Per the North American Research Committee on Multiple Sclerosis, a survey was conducted on spasticity prevalence and results show 84% have some degree of spasticity from mild to incapacitating. Spasticity pathophysiology is complex and not completely understood with higher levels of incapacitating spasticity reported in this survey by those who were male, disabled and unemployed, indicating that psychosocial and subjective variables are significant. The pathophysiology currently best understood demonstrates an imbalance between inhibitory dorsal reticulospinal tract (RST) fibers and excitatory bulbopontine tegmentum. RST neurons receive direct somatic, vestibular, tectal, cerebellar and motor excitatory input and are scattered in the ventral and lateral spinal cord columns intermingled with propriospinal fibers. The peripheral Golgi tendon organ of muscle tendon and muscle spindle intrafusal fibers ubiquitous throughout the musculoskeletal system have direct monosynaptic connection to these central nervous system propriospinal fibers and heavily influence the degree of spasticity and overactive stretch reflexes.

Those who deal with all levels of spasticity use compensatory movement strategies causing altered arthrokinematics and have loss of strength, balance and efficient muscle use with postural changes. Spasticity management has been studied and treated from a pharmaceutical standpoint with some improvements but often side effects including fatigue, muscle weakness and cognition limit dosing in oral Baclofen, Dantrolene Sodium, Tizanidine and Benzodiazepines. Marijuana especially in form of cannabinoids shows mixed evidence for spasticity improvement and is a growing area of interest. There is a growing CBD interest in the MS population due to known reduction of CNS neurodegeneration in animal MS studies and no significant negative side effects with possible mild to moderate improvement in spasticity levels. Therapy interventions offered include frequent stretching especially of muscles that cross two joints including lumbricals, hamstrings, gastrocnemius and iliopsoas; light stroking over lower limbs demonstrated a 30% decrease in H-reflex amplitude lasting even 30 minutes after treatment; muscle cooling was shown to reduce muscle stretch activity and clonus; Armutlu et al. Reported significant reduction in plantar flexor spasticity in 10 patients with MS using high-frequency (100Hz) TENS for 20min daily for 4 weeks. Reduction noted on Modified Ashworth Scale (MAS), electrophysiologic measurements and the AI; and serial casting performed over a 9-day period with cast changes every 3 days demonstrated reduced spasticity levels.

The NeuFit company offers a Neubie EMS product with a direct current using high fidelity audio equipment to decrease intensity of the treatment noxious stimulus and protect skin integrity from burns or intolerable pain. This system uses an exponential wave pattern to mimic the natural pattern neurologically to lengthen fibers of the sarcomere and engage force velocity of muscle with minimized protective co-contraction of nearby muscle groups9. The golgi tendon and muscle spindles code for joint position and muscle/tendon stretch with 66% of fibers being intrafusal. Impacting these structures has direct impact on reticulospinal tract (RST) fibers and proprioceptive central fibers modulation of levels of spasticity. However, finding effective means to impact these areas is difficult. The Neubie direct current is designed to improve positioning of these stretch receptors. As discussed within the paper hypothesis, the theory is that this may improve spasticity levels as well as agonist strength enough to create long term, significant functional improvement.

Dr. Terry Wahls who has MS and has studied and marketed a protocol for MS treatment, promotes this product and has a home unit she uses daily to control her own MS symptoms and gain strength. Currently there is no research study conducted on the effects of the Neubie direct current treatment combined with exercise and ramifications of spasticity in multiple sclerosis. There have been only a few studies conducted with quantitative spasticity measures mostly with FES and NMES targeting tibialis anterior and quadriceps to lessen plantar flexor spasticity in spinal cord injury (SCI) and hemiplegia. In the SCI study Mirbagheri et al. observed decreases in intrinsic and reflex dynamic stiffness in all 4 subjects studied over a 16-month period. Robinson et al. stimulated quadriceps muscle pulse duration 500, 20 Hz and amplitude of 100 with spasticity quantitatively reduced immediately after stimulation but return of baseline spasticity level when measured 24 hours later. Levin and Hui-Chan assessed sensory level stimulation of the common peroneal nerve for a total of 15, 60 min sessions for 3 weeks in people with hemiplegia using pulse duration 125 continuously at 99Hz and observed inhibition of H-reflex at soleus, increase in dorsiflexion voluntary force and reductions in stretch reflex at triceps surae. The NeuFit method of treatment allows the recipient to voluntarily concentrically or eccentrically activate muscles while receiving the direct current passive eccentric input. In order to assess the feasibility of this papers' hypothesis the investigators will perform a pilot study of 4-6 individuals with MS in the greater Denver metro area.

ELIGIBILITY:
Inclusion Criteria:

1. Greater than 18 years old (no upper age limit)
2. Physician diagnosed MS (As stated in Rooney S, et al. Disabil Rehabil. 2019, stage of MS did not impact individuals from making neuromuscular or functional gains. All stages of MS will be eligible)
3. Physician clearance to participate
4. Unable to ambulate more than 70 feet at a time and unable to ambulate outside the home, with use of manual chair or power chair as mobility source >= 50% of the time.
5. BLE MMT in hips, knees and ankles <=3/5
6. Modified Ashworth assessed spasticity levels 1-4

Exclusion Criteria:

1. Co-morbidities in cardiovascular disease (myocardial infarction in past 1-year, unstable angina, CHF, h/o arrythmia, h/o CVA or TIA in past year, uncontrolled hypertension)
2. History of epileptic seizures
3. Lower Motor Neuron disease
4. Existing pacemaker, defibrillator or other implanted device (other than baclofen pump)
5. Unstable long bone fractures of lower limb or trunk
6. Allergies to surface electrodes or conductive gel
7. Pregnancy or actively seeking to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-06-20 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Ellerbusch, DPT, Principal Investigator — CommonSpirit Health
Locations (1):
- Centura Health at Home, Littleton, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Backus D, Burdett B, Hawkins L, Manella C, McCully KK, Sweatman M. Outcomes After Functional Electrical Stimulation Cycle Training in Individuals with Multiple Sclerosis Who Are Nonambulatory. Int J MS Care. 2017 May-Jun;19(3):113-121. doi: 10.7224/1537-2073.2015-036. PMID 28603459
- [Background] Etoom M, Khraiwesh Y, Lena F, Hawamdeh M, Hawamdeh Z, Centonze D, Foti C. Effectiveness of Physiotherapy Interventions on Spasticity in People With Multiple Sclerosis: A Systematic Review and Meta-Analysis. Am J Phys Med Rehabil. 2018 Nov;97(11):793-807. doi: 10.1097/PHM.0000000000000970. PMID 29794531
- [Background] Wahls TL, Reese D, Kaplan D, Darling WG. Rehabilitation with neuromuscular electrical stimulation leads to functional gains in ambulation in patients with secondary progressive and primary progressive multiple sclerosis: a case series report. J Altern Complement Med. 2010 Dec;16(12):1343-9. doi: 10.1089/acm.2010.0080. PMID 21138391
- [Background] Szecsi J, Schlick C, Schiller M, Pollmann W, Koenig N, Straube A. Functional electrical stimulation-assisted cycling of patients with multiple sclerosis: biomechanical and functional outcome--a pilot study. J Rehabil Med. 2009 Jul;41(8):674-80. doi: 10.2340/16501977-0397. PMID 19565162
- [Background] Mills PB, Dossa F. Transcutaneous Electrical Nerve Stimulation for Management of Limb Spasticity: A Systematic Review. Am J Phys Med Rehabil. 2016 Apr;95(4):309-18. doi: 10.1097/PHM.0000000000000437. PMID 26829077
- [Background] Meseguer-Henarejos AB, Sanchez-Meca J, Lopez-Pina JA, Carles-Hernandez R. Inter- and intra-rater reliability of the Modified Ashworth Scale: a systematic review and meta-analysis. Eur J Phys Rehabil Med. 2018 Aug;54(4):576-590. doi: 10.23736/S1973-9087.17.04796-7. Epub 2017 Sep 13. PMID 28901119

RESULTS

PARTICIPANT FLOW:
Groups:
- Neubie Treatment: Outcome measures will be collected at the beginning and end of study.
  1. Manual activations to underactive, spastic or limited in sensory muscles/regions
  2. Neubie Mapping mode scanning process to scan for 1) spots that stimulate movement they couldn't do before per initial assessment, 2) spots that allow movement which is a greater range than available before per initial assessment, 3) spots that lead to decreased spasticity, and 4) diminished sensation areas - drive signal to increase sensory nerves and become metabolically active.
  3. Train using physical therapy exercises with Neubie in training mode and Hz current adjusted for tolerance (perceived 7/10) and ability to work through or decrease spasticity in (500 Hz) in the areas which show spasticity, contraction, are dead/diminished sensation, and hot spots.
  Neubie: The Neubie is a direct current neuromuscular electrical stimulation device. This system uses an exponential wave pattern to mimic the natural pattern neurologically to lengthen fibers of the sarcomere and engage force velocity of muscle with minimized protective co-contraction of nearby muscle groups. The golgi tendon and muscle spindles code for joint position and muscle/tendon stretch with 66% of fibers being intrafusal. Impacting these structures has direct impact on reticulospinal tract fibers and proprioceptive central fibers modulation of levels of spasticity. The Neubie direct current is designed to improve positioning of these stretch receptors.
Period: Overall Study
Arm/Group | Neubie Treatment
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Neubie Treatment: All participants in this study will participate in intervention treatment with the Neubie for 6 weeks. Outcome measures objective and subjective will be collected at the beginning and end of the study. The treatments will include:
  1. Manual activations to underactive, spastic or limited in sensory muscles/regions
  2. Neubie Mapping mode scanning process to scan for 1) spots that stimulate movement they couldn't do before per initial assessment, 2) spots that allow movement which is a greater range than available before per initial assessment, 3) spots that lead to decreased spasticity, and 4) diminished sensation areas - drive signal to increase sensory nerves and become metabolically active.
  3. Train using physical therapy exercises with Neubie in training mode and Hz current adjusted for tolerance (perceived 7/10) and ability to work through or decrease spasticity in (500 Hz) in the areas which show spasticity, contraction, are dead/diminished sensation, and hot spots.
Arm/Group | Neubie Treatment
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Expanded Disability Status Score
Description: The Expanded Disability Status Scale (EDSS) is a method of quantifying disability in multiple sclerosis and monitoring changes in the level of disability over time. It is widely used in clinical trials and in the assessment of people with MS.The EDSS scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability. Scoring is based on an examination by a neurologist. The neurologist did not measure any change in EDSS score for any of the 7 study subjects from her first assessment to her final second assessment.
Time Frame: Baseline, Pre-intervention
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Neubie Treatment
Number analyzed (Participants) | 7
score on a scale | 6.8 (0.8)

2. Primary Outcome: Expanded Disability Status Score
Description: as for outcome 1
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neubie Treatment
Number analyzed (Participants) | 7
score on a scale | 6.8 (0.8)

3. Primary Outcome: 12 Item MS Walking Scale
Description: The Multiple Sclerosis Walking Scale is a self-assessment scale which measures the impact of MS on walking. It consists of 12 questions concerning the limitations to walking due to MS. Each item can be answered with 5 options, with 1 meaning no limitation and 5 extreme limitation. A total score can be generated and transformed to a 0 to 100 scale by subtracting the minimum score possible (12) from the patient's score, dividing by the maximum score possible minus the minimum possible (60-12 or 48), and multiplying the result by 100. Walking improvement on the MSWS-12 is indicated by negative change scores.
Time Frame: Baseline, Pre-intervention
Measure: Mean (Standard Deviation); unit: percentage of a score on a scale
Groups:
- Neubie Treatment: Adult individuals with confirmed diagnosis of Multiple Sclerosis. Summarize inclusion and exclusion criteria...
Arm/Group | Neubie Treatment
Number analyzed (Participants) | 7
percentage of a score on a scale | 0.89 (0.14)

4. Primary Outcome: 12 Item MS Walking Scale
Description: as for outcome 3
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: percentage of a score on a scale
Arm/Group | Neubie Treatment
Number analyzed (Participants) | 7
percentage of a score on a scale | 0.7 (0.28)

5. Primary Outcome: Manual Muscle Test
Description: A standardized set of assessments that measure strength. Scores are provided for each assessed muscle or muscle group individually in a scale from 0 to 5, in which 0 means no palpable muscle contraction, and 5 means a full range of motion capable of resisting 5 pounds of pressure. This scale of 5 includes values of (-) and (+) for each number which equals a total of 12. Data is entered on a 12-point scale here per requirements in data entry per clinical trials.
Time Frame: Baseline, Pre-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neubie Treatment
Number analyzed (Participants) | 7
score on a scale
  Psoas right | 4 (2)
  Psoas left | 4 (3)
  rectus abdominus | 4 (2)
  quadratus lumborum right | 4 (1)
  quadratus lumborum left | 5 (2)
  rectus femoris right | 4 (2)
  rectus femoris left | 5 (2)
  vastus lateralis and medialis right | 6 (4)
  vastus lateralis and medialis left | 6 (3)
  gluteus medius right | 5 (2)
  gluteus medius left | 5 (3)
  adductor group right | 6 (2)
  adductor group left | 6 (2)
  tibialis anterior right | 5 (4)
  tibialis anterior left | 6 (4)
  fibularii right | 6 (4)
  fibularii left | 6 (4)
  lumbar extension | 8 (3)
  gluteus maximus right | 4 (3)
  gluteus maximus left | 4 (2)

6. Primary Outcome: Manual Muscle Test
Description: as for outcome 5
Time Frame: 3 week measurement
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neubie Treatment
Number analyzed (Participants) | 7
units on a scale
  Psoas right | 3 (2)
  Psoas left | 4 (2)
  rectus abdominus | 4 (1)
  quadratus lumborum right | 5 (3)
  quadratus lumborum left | 4 (2)
  rectus femoris right | 3 (2)
  rectus femoris left | 4 (2)
  vastus lateralis and vastus medialis left | 6 (3)
  vastus lateralis and vastus medialis right | 7 (3)
  gluteus medius right | 5 (2)
  gluteus medius left | 5 (2)
  adductor group right | 6 (1)
  adductor group left | 6 (1)
  tibialis anterior right | 3 (3)
  tibialis anterior left | 5 (3)
  fibularis right | 3 (3)
  fibularis left | 5 (3)
  lumbar extension | 7 (4)
  gluteus maximus right | 4 (2)
  gluteus maxiums left | 4 (2)

7. Primary Outcome: Manual Muscle Test
Description: as for outcome 5
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neubie Treatment
Number analyzed (Participants) | 7
units on a scale
  psoas right | 4 (2)
  rectus abdominus | 5 (1)
  rectus femoris right | 5 (1)
  rectus femoris left | 5 (3)
  gluteus maxiumus left | 5 (3)
  biceps femoris right | 6 (2)
  gluteus maximus right | 6 (3)
  psoas left | 6 (2)
  biceps femoris left | 6 (2)
  tibialis anterior right | 6 (4)
  quadratus lumborum left | 3 (2)
  gluteus medius left | 6 (3)
  gluteus medius right | 7 (2)
  quadratus lumborum right | 7 (2)
  tibialis anterior left | 7 (3)
  vastus lateralis/medialis right | 8 (3)
  hip adductor group right | 8 (2)
  lumbar extension bilateral | 8 (3)
  vastus lateralis/medialis left | 9 (4)
  hip adductor group left | 9 (2)

8. Primary Outcome: Timed 25 Foot Walk Test (T25FW)
Description: The T25FW is a clinical tool that evaluates patients for quantitative mobility and leg function performance test in time, 25 foot walk.
Time Frame: Baseline, Pre-intervention
Measure: Mean (Standard Deviation); unit: units on a scale (seconds)
Arm/Group | Neubie Treatment
Number analyzed (Participants) | 7
units on a scale (seconds) | 21.4 (5.2)

9. Primary Outcome: Multiple Sclerosis Impact Scale (MSIS-29)
Description: The Multiple sclerosis impact scale 29 (MSIS-29) is a 29-item assessment combining questions about the physical and psychological impact of the participant's condition on daily living. All items have Likert style response options that go from 1 (not at all) to 5 (extremely), where a total score of 145 indicates greater impact of disease on daily function (worse health), and the lower the score (The closer it is to 29), the smaller the impact of multiple sclerosis on the participant's daily function.
Time Frame: baseline, pre-intervention
Measure: Mean (Standard Deviation); unit: percentage of a score on a scale
Arm/Group | Neubie Treatment
Number analyzed (Participants) | 7
percentage of a score on a scale | 97.3 (25.2)

10. Primary Outcome: Timed 25 Foot Walk Test (T25FW)
Description: The T25FW is a clinical tool that evaluates patients for quantitative mobility and leg function performance test in time, 25-foot walk measured in seconds. Higher second measures are slower and considered "worse" while lower second measures are faster and considered "better".
Time Frame: 3 week
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Neubie Treatment
Number analyzed (Participants) | 7
seconds | 20.7 (5.9)

11. Primary Outcome: Timed 25 Foot Walk Test (T25FW)
Description: as for outcome 10
Time Frame: 6 week
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Neubie Treatment
Number analyzed (Participants) | 7
seconds | 15 (1.3)

12. Primary Outcome: Multiple Sclerosis Impact Scale (MSIS-29)
Description: as for outcome 9
Time Frame: 6 week
Measure: Mean (Standard Deviation); unit: percentage of a score on a scale
Arm/Group | Neubie Treatment
Number analyzed (Participants) | 7
percentage of a score on a scale | 85 (20.2)

13. Primary Outcome: Modified Ashworth Test
Description: The Modified Ashworth Test is measured on a 5-point scale used to assess spasticity by grading the resistance encountered during passive muscle stretching. The assessor rates the perceived amount of resistance or tone encountered during the range of motion.
  0=no tone detected
  1+ = tone able to move through for less than half the range 2=tone able to move through for more than half the range 3=significant resistance to movement for entire range but able to break tone 4=completely rigid and unable to move limb
Time Frame: Baseline, pre-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Neubie Treatment: Adult individuals with confirmed diagnosis of Multiple Sclerosis.
Arm/Group | Neubie Treatment
Number analyzed (Participants) | 7
units on a scale
  ankle dorsiflexion left | 0 (0)
  knee extension left | 1 (1)
  ankle dorsiflexion right | 0 (0)
  ankle plantarflexion right | 3 (1)
  knee extension right | 1 (1)
  ankle plantarflexion left | 2 (1)
  hip extension left | 1 (1)
  hip flexion left | 0 (1)
  knee flexion left | 1 (1)
  hip extension right | 1 (1)
  hip flexion right | 0 (0)
  knee flexion right | 1 (1)

14. Primary Outcome: Modified Ashworth Test
Description: as for outcome 13
Time Frame: 6 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neubie Treatment
Number analyzed (Participants) | 7
units on a scale
  ankle dorsiflexion left | 0 (0)
  knee extension left | 1 (1)
  ankle dorsiflexion right | 0 (0)
  ankle plantarflexion right | 2 (1)
  knee extension right | 1 (1)
  ankle plantarflexion left | 2 (1)
  hip extension left | 1 (1)
  hip flexion left | 0 (0)
  knee flexion left | 0 (1)
  hip extension right | 0 (0)
  hip flexion right | 0 (0)
  knee flexion right | 1 (1)

ADVERSE EVENTS:
Time Frame: 1 day
Description: Adverse event collection match the clinicaltrials.gov definitions and procedures.
Groups:
- NeuBie Treatment: The 7 subjects with Multiple Sclerosis participating in this clinical trial.
Arm/Group | NeuBie Treatment
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NeuBie Treatment (N=7)
Fatigue (General disorders) | 1 (1) — The patient presented with fatigue and symptoms suggestive of urinary tract infection which limited her capacity to tolerate the study required ambulatory testing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-05-24): https://cdn.clinicaltrials.gov/large-docs/38/NCT04942938/Prot_001.pdf
  • Statistical Analysis Plan (2022-07-21): https://cdn.clinicaltrials.gov/large-docs/38/NCT04942938/SAP_002.pdf